CLINICAL TRIAL: NCT01580904
Title: Popular Pharmacy of Brazil: Impact of Pharmaceutical Care in Diabetics Patients
Brief Title: Impact of Pharmaceutical Care in Diabetics Patients
Acronym: IPCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual da Paraiba (Other)
Collaborators: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Patrícia Trindade Costa Paulo, Impact of Pharmaceutical Care in Diabetics Patients: Clinical Trial Randomized, Universidade Estadual da Paraiba
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UEParaiba
Record Dates: First submitted 2012-04-11; First posted 2012-04-19 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Pharmaceutical Care; Diabetics patients; Clinical trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): Patients will not be followed by the pharmacist.
- Intervention group (Experimental): Patients will be followed by the pharmacist by Pharmacotherapeutic monitoring and dosing parameters such as glucose and glycated hemoglobin.
  Intervention: Pharmaceutical Care
  Interventions: Behavioral: Intervention: Pharmaceutical Care

INTERVENTIONS:
Behavioral: Intervention: Pharmaceutical Care — Patients will be followed by the pharmacist by the Pharmaceutical Care Practice
  Arms: Intervention group

SUMMARY:
The monitoring of diabetics by the pharmacist may contribute to the effectiveness of drug treatment and to improve their quality of life. This study will measure the impact of pharmacotherapeutic follow-up in diabetic patients. This will be a clinical trial, single blind, controlled, randomized, conducted in two units of pharmacies in Brazil. Only in the intervention group will be held the pharmacotherapeutic follow using a methodology called the practice of pharmaceutical care, which identifies and resolves problems related to drugs. The primary outcome is glycated hemoglobin, and secondary outcomes are baseline glucose, total cholesterol and its fractions (for example LDL), all these measures will be made in the intervention group and control group. Patients will be followed for 24 weeks, and the outcomes will be assessed up to 24 weeks. There will be a confidence interval of 95% and a significance of p <0.05, and will use the Student t test, chi-square analysis of variance (ANOVA) and others if necessary. Expects good results and serve as a model for other researchers.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria:

* patients aged 30 years,
* diagnosed with type 2 diabetes,
* to make use of oral antidiabetic agents with or without insulin

Exclusion Criteria:

those who had infectious diseases during the research

* missed three consecutive interviews,
* suspended the hypoglycemic drug and medical order

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivonete A. Doutorado, Study Director — Universidade Federal do Rio Grande do Norte
Locations (1):
- Universidade Estadual da Paraíba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell B, Armour C, Lee M, Song YJ, Stewart K, Peterson G, Hughes J, Smith L, Krass I. Diabetes Medication Assistance Service: the pharmacist's role in supporting patient self-management of type 2 diabetes (T2DM) in Australia. Patient Educ Couns. 2011 Jun;83(3):288-94. doi: 10.1016/j.pec.2011.04.027. Epub 2011 May 26. PMID 21616627
- See also: A journal that has a lot of research on this topic — http://www.pharmacypractice.org/
- See also: An interesting article on this topic — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2387287/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2009 to December 2011.Medical clinic
Pre-assignment Details: The exclusion criteria were (i) to have an infectious disease during the study, (ii) to miss three consecutive appointments, (iii) to stop the use of the hypoglycemic drugs by order of the doctor, and (iv) to deny the acceptance of the term of free and informed consent (TFIC).
Groups:
- Intervention Group: Patients will be followed by the pharmacist.
  Intervention: Pharmaceutical Care : Patients will be followed by the pharmacist by the Pharmaceutical Care Practice
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 51 | 49
Completed | 47 | 42
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 47 | 42 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 30 | 67
  >=65 years | 10 | 12 | 22
Gender [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  Brazil | 47 | 42 | 89

OUTCOME MEASURES:

1. Primary Outcome: Glycated Hemoglobin
Description: average glycated hemoglobin over 24 weeks
Time Frame: Up to 24 weeks
Population: Data are glycated hemoglobin means of all patients per group.
Measure: Mean (Standard Deviation); unit: percent (%)
Groups:
- Intervention Group: Patients will be followed by the pharmacist.
  Intervention: Pharmaceutical Care: Patients will be followed by the pharmacist by the Pharmaceutical Care Practice
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 42 | 47
percent (%) | 7.2 (1.5) | 7.1 (1.7)

2. Primary Outcome: Fasting Glycemia
Description: average fasting glycemia over 24 weeks
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Intervention Group: Patients will be followed by the pharmacist by Pharmacotherapeutic monitoring and dosing parameters such as glucose and glycated hemoglobin.
  Intervention: Pharmaceutical Care
  Intervention: Pharmaceutical Care: Patients will be followed by the pharmacist by the Pharmaceutical Care Practice
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 42 | 47
mg/dL | 157.7 (43.1) | 159.3 (56.7)

3. Secondary Outcome: Total Cholesterol
Description: average total cholesterol over 24 weeks
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 42 | 47
mg/dL | 209.9 (42.8) | 191.1 (36.5)

4. Secondary Outcome: LDL Cholesterol
Description: average LDL cholesterol over 24 weeks
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 42 | 47
mg/dL | 131.0 (33.0) | 110.8 (32.4)

ADVERSE EVENTS:
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 31/42 | 34/47
Other Adverse Events (participants affected / at risk) | 30/42 | 32/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=42) | Intervention Group (N=47)
Stomach pain (Gastrointestinal disorders) | 31 | 34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=42) | Intervention Group (N=47)
Queasiness (Cardiac disorders) | 30 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes